## **Protocol**

Title: Myo-inositol in prevention of gestational diabetes mellitus in China

RCT Number: Date: Feb 4<sup>th</sup>, 2021



## Planned Analysis

- 1) Chi square test and t test are used to compare the basic information of the subjects.
- 2) T test is used to compare the results of OGTT between the intervention group and the control group
- 3) Chi square test is used to analyze the incidences of secondary outcomes (such as cesarean section rate, weight gain, macrosomia etc) between the intervention group and the control group
- 4) Logistic regression and linear regression analysis were used to calculate the association between inositol intake and other confounding factors (such as age, BMI, etc.).